CLINICAL TRIAL: NCT03814395
Title: Peking University Birth Cohort in Tongzhou
Acronym: PKUBC-T
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Hai-Jun Wang, Prof., Peking University
Other Study IDs: NNSF81703240; 81703240 (Other Grant/Funding Number: The National Natural Science Fund)
Record Dates: First submitted 2019-01-16; First posted 2019-01-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Health Problems in Pregnancy; Pregnancy Outcomes; Gestational Diabetes; Gestational Hypertension; Preterm Birth; Obesity; Mother-Infant Interaction; Child Development; Anemia
MeSH Terms: conditions — Diabetes, Gestational; Hypertension, Pregnancy-Induced; Premature Birth; Obesity; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During pregnancy: maternal blood. At delivery: cord blood，umbilical cord and placenta. During childhood: blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group: Group with environmental, nutritional or lifestyle exposures
  Interventions: Other: No intervention
- Non-exposed group: Group without any environmental, nutritional and lifestyle exposures

INTERVENTIONS:
Other: No intervention — This is an observational study without any intervention
  Groups: Exposure group

SUMMARY:
The PKUBC-T is a prospective cohort study carried out in Tongzhou district of Beijing, China. The primary aim of this study is to investigate the short-term and long-term effects of pre-pregnant and prenatal exposure on maternal and child health. Data are collected regarding environmental, nutritional and lifestyle exposures as well as short-term and long-term health outcomes of mothers and their children from birth to 6 years old. Biological samples including blood and tissue samples are also collected from mothers and their children.

DETAILED DESCRIPTION:
Maternal and child health is of great concern globally. Early life phase of a fetus and infant is a critical period for the development of health and disease in the whole life. Exposure of negative environmental, nutritional and lifestyle factors in pregnant women during this period can have adverse effects on fetal and infant. In addition, for mothers, complications during pregnancy could also have a negative effect on long-term health of mothers, such as diabetes, hypertension. Thus, the Peking University Birth Cohort in Tongzhou is primarily aimed to investigate the short-term and long-term effects of pre-pregnant and prenatal exposure on maternal and child health. Data are collected regarding environmental, nutritional and lifestyle exposures as well as short-term and long-term health outcomes of mothers and their children from birth to 6 years old. Biological samples including blood and tissue samples are also collected from mothers and their children.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women, <14 gestational weeks
2. Resided in Tongzhou in the past half years and have no plan to move out after delivery
3. Pregnant women who plan to have antenatal care and delivery in Tongzhou maternal&Child Hospital.
4. Pregnant women who is willing to participate in this study with informed consent

Exclusion Criteria:

Pregnant women have chronic disease before pregnancy, including diabetes，hypertension, liver disease and kidney disease.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women and their children in Tongzhou, China
Sampling Method: Non-Probability Sample
Enrollment: 5426 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with pregnancy complications | At delivery
  Including gestational diabetes, gestational hypertension, anemia, and hypothyroidism during pregnancy
Numbers of participants with adverse pregnancy outcomes | At delivery
  Including preterm birth, low birth weight, macrosomia, abortion, stillbirth, and birth defects.

SECONDARY OUTCOMES:
Weight in kilogram changes during childhood | At birth and age at 6 weeks, 3 months, 6 months, 8 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years, 4 years, 5 years and 6 years
  Measured by health professionals in clinic
Height in centimeter changes during childhood | At birth and age at 6 weeks, 3 months, 6 months, 8 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years, 4 years, 5 years and 6 years
  Measured by health professionals in clinic
Early Child development 1 | Age at 6 weeks and 3 years
  Measured by Ages&Stages Questionnaires (ASQ).There are 6 questions in each of 5 domains of development: communication, gross motor, fine motor, problem-solving skills, and adaptive skills. Each question is given a 10 (yes), 5 (sometimes), or 0 (not yet) score according to the parents' answers. The sum scores (range from 0 to 300) and scores for each domain (range from 0 to 60) are calculated. Chinese norms are available for each domain, and any domain screened <2 SDs below the mean is considered a positive screening. A higher ASQ score means better development.
Early Child development 2 | Age at 8-12 months
  Measured by Denver Developmental Screening Test (DDST). DDST comprises 125 test items grouped into four domains of child development: 25 personal-social (PS), 29 fine motor (FM), 39 language (LA) and 32 gross motor (GM). These test items are administered using a bell, glass bottle, set of 10 blocks, rattle, pencil, tennis ball, yarn, raisins, cup, white doll, white paper, and baby bottle. A child's raw score on each test item is marked as tested pass, failure, refusal, or no opportunity. The result of the test is labeled as "normal," "suspect" or "abnormal". Normal development means that there is no delay or at the maximum one warning. Abnormal development means that there is one or more than one delay situation. Suspicious development means that it is a situation involving one delay, one delay and one warning or two or more than two warnings. The number of children with normal, suspect or abnormal development is calculated.
Incidence of diabetes mellitus in women | 6 weeks after delivery and 3 years after delivery
  Measured by health professionals in clinic
Incidence of hypertension in women | 6 weeks after delivery and 3 years after delivery
  Measured by health professionals in clinic
Incidence of child overweight and obesity | Age at 6 weeks, 3 months, 6 months, 8 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years, 4 years, 5 years and 6 years
  Measured by health professionals in clinic
The proportion of children with warning signs | Age at 3 months, 6 months, 8 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years, 4 years, 5 years and 6 years
  Measured by warning signs screening
Fetal Biparietal Diameter | At 20-24 gestational week, 30-32 gestational week and 37-41 gestational week.
  Measured by health professionals in clinic with ultrasound
Fetal Head Circumference | At 20-24 gestational week, 30-32 gestational week and 37-41 gestational week.
  Measured by health professionals in clinic with ultrasound
Fetal Abdominal Circumference | At 20-24 gestational week, 30-32 gestational week and 37-41 gestational week.
  Measured by health professionals in clinic with ultrasound
Fetal Femur Length | At 20-24 gestational week, 30-32 gestational week and 37-41 gestational week.
  Measured by health professionals in clinic with ultrasound
Fetal Humerus Length | At 20-24 gestational week, 30-32 gestational week and 37-41 gestational week.
  Measured by health professionals in clinic with ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Haijun Wang, Ph.D, Principal Investigator — Peking University
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jin C, Lin L, Han N, Zhao Z, Liu Z, Luo S, Xu X, Liu J, Wang H. Effects of dynamic change in fetuin-A levels from the first to the second trimester on insulin resistance and gestational diabetes mellitus: a nested case-control study. BMJ Open Diabetes Res Care. 2020 Jan;8(1):e000802. doi: 10.1136/bmjdrc-2019-000802. PMID 31958310